| <b>Document Type:</b> | Statistical Analysis Plan |
|---|---|
| Official Title: | A 2-stage, Lead-In and Randomized, Phase 2, Open-label study of Darolutamide versus Enzalutamide as Monotherapy on Testosterone Levels Change in Men with Hormone-Naïve Prostate Cancer (ARAMON) |
| NCT Number: | NCT05526248 |
| <b>Document Date:</b> | 06 MAR 2024 |

#### ARAMON V3.0



Page: 1 of

# **Title Page**

**Protocol Title:** A 2-stage, Lead-in and Randomized, Phase 2, Open-label study of Darolutamide versus Enzalutamide as Monotherapy on Testosterone Levels Change in Men with Hormone-Naïve Prostate Cancer (ARAMON)

**Protocol Number:** BAY 1841788 / 21953

Compound Number: BAY 1841788 / Darolutamide

**Short Title:** ARAMON: Evaluation of darolutamide versus enzalutamide monotherapy in

men with hormone naïve Prostate Cancer

Acronym: ARAMON

**Sponsor Name:** Bayer HealthCare Pharmaceuticals, Inc.,

**Legal Registered Address:** 100 Bayer Boulevard, P.O. Box 915, Whippany, NJ 07981-0915, USA

#### **Regulatory Agency Identifier Number(s):**

**Registry** ID

**IND** 114769

NCT 05526248

**Date:** 06 MAR 2024

Version: 3.0

#### Confidential

The information provided in this document is strictly confidential and is intended solely for the performance of the clinical investigation. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the clinical investigation or its use for any other purpose without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) may not be displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

This Statistical Analysis Plan is produced on a word-processing system and bears no signatures. The approval of the Statistical Analysis Plan is documented in a separate signature document.

# **Table of Contents**

| Title Page 1 | |
|-------------------------------------------|----|
| Table of Contents | 2 |
| Γable of Tables | |
| Table of Figures | 3 |
| Version History | 4 |
| 1. Introduction | |
| 1.1. Objectives, Endpoints, and Estimands | |
| 1.2. Study Design | |
| 1.2.1 Overall Design | |
| 1.2.1.1 Screening period | |
| 1.2.1.2 Treatment period | |
| 1.2.1.3 Active Follow–up period | |
| 1.2.2 Participant completion of study | |
| 1.2.3 End of Study Definition | 9 |
| 2. Statistical Hypotheses | 10 |
| 2.1. Multiplicity Adjustment | |
| 3. Analysis Sets | 11 |
| 4. Statistical Analyses | 12 |
| 4.1. General Considerations | |
| 4.1.1 Analysis junctures | 12 |
| 4.1.2 Handling missing data | 12 |
| 4.1.3 Data rules | |
| 4.2. Primary Endpoint Analysis | |
| 4.2.1 Main Analytical Approach | |
| 4.2.1.1 Lead-in Phase | |
| 4.2.1.2 Randomized Phase | |
| 4.3. Secondary Endpoint Analysis | |
| 4.3.1 Main Analytical Approach | |
| 4.3.1.1 Lead-in Phase | |
| 4.3.1.2 Randomized Phase | |
| 4.5. Safety Analyses | |
| 4.5.1 Extent of Exposure | |
| 4.5.2 Adverse Events | |
| 4.6. Other Analyses | |
| 4.6.1 Lead-in Phase Analyses | |
| 4.6.2 Subgroup Analyses | |
| 4.7. Interim Analyses | |
| 4.8. Changes to Protocol-planned Analyses | |
| 5. Sample Size Determination | |
| Lead-in Phase | |
| Randomized Phase | 20 |
| 6. Supporting Documentation | 21 |

# Statistical Analysis Plan 1841788 / 21953

ARAMON V3.0 

| 6.1. | Population Characteristics | 21 |
|---|---|---|
| 6.1.1 | Disposition of participants | 21 |
| 6.1.2 | Demographics and baseline characteristics | 21 |
| 6.1.3 | Prior anti-cancer therapies | 22 |
| 6.1.4 | Important protocol deviations | 22 |
| | x 1: Imputation rule for partial missing dates | |
| Appendi | x 2: Scoring procedures for FACT-P | 23 |
| Appendi | x 3: Scoring for PROMIS | 25 |
| Appendi | x 4: Randomized phase primary endpoint analysis for natural logarithm transformed Testosterone | |
| Appendi | x 5: Lead-in phase analysis for natural logarithm transformed Testosterone and other | r |
| | endpoints using the log transformation | 27 |
| Appendi | x 6: Randomized phase analysis for natural logarithm transformed Testosterone and | |
| | other endpoints using the log transformation | 28 |
| Appendi | x 7: List of Abbreviations | 30 |
| Table o | of Tables | |
| Table 1- | 1: Lead-in phase objectives and Endpoints | . 7 |
| | 2: Randomized Phase Objectives and Endpoints | |
| | 1: Populations for analyses: Lead-in phase | |
| | 2: Populations for analyses: Randomized Phase | |
| Table o | of Figures | |
| Figure 1 | -1: Overall Design | . 8 |

ARAMON V3.0 

# **Version History**

This Statistical Analysis Plan (SAP) for Study ARAMON is based on the protocol Version 2.0 dated 10 AUG 2023.

| SAP Version | Date | Rationale | |
|---|---|---|---|
| 1.0 | 31 AUG 2022 | Not applicable | Original version |
| 2.0 | 18 JAN 2024 | Section 1.1: Revise endpoint language in table 1-1 and 1-2. | Align with protocol v2.0 |
| | | Section 1.1: Add fasting insulin as an endpoint and footnotes updated in table 1-2. | Align with protocol v2.0 |
| | | Section 1.1: Remove Week 12 from testosterone secondary endpoint in tables 1-1 and 1-2. | Align with protocol v2.0 and remove redundancy with primary endpoint |
| | | Section 1.2: Add details on data cut type used for the analysis | Clarification on what data to be used for the analysis |
| | | Section 1.2.1: Add footnote to Figure 1-1 | Align with protocol v2.0 |
| | | Section 1.2.1.2: Add EOT treatment visit details. | Align with protocol v2.0 |
| | | Section 1.2.1.3: Revise Active follow-up period definition. | Align with protocol v2.0 |
| | | Section 3: Change 'met all inclusion exclusion criteria' to 'met all inclusion and none of the exclusion criteria' | Align with protocol v2.0 |
| | | Section 4.1.3: Remove 'within +/- 7 days of scheduled date' | Account for baseline measures done outside the window |
| | | Section 4.1.3: Clarify the nearest measure prior to the study drug administration date will be used for baseline | To include the baseline measures recorded in the 'Unscheduled' visit CRF pages |
| | | Section 4.1.3: Revise the logic to choose the measurement for the analysis | Remove ambiguity around 'scheduled date' and to include 'unscheduled' pos baseline measurement incase scheduled visits do not exist |
| | | Section 4.2.1: Remove 'darolutamide' from the primary analysis timepoint for randomized phase | Align with protocol v2.0 that last participant could be on either arm in randomized phase |
| | | Section 4.3.1.1 Change 'absolute' PSA response to 'Undetectable' PSA response, and 50% and 90% 'relative' PSA response to PSA50, PSA90. | Align with terminologies commonly used in other literature |
| | | Section 4.3.1.1 Remove relative 30% PSA response (PSA30) | To focus on PSA50 and PSA90 since response rate in mHSPC is very high |
| | | Section 4.3.1.1 Add 0.2 ng/mL detection limit value to PSA response rates definitions | Clarify detection limit |
| | | Section 4.3.1.1 Add Breast enlargement, Breast | Summarize all AEs classified as feminizing side-effects |
| | | mass, Breast swelling in gynecomastia Section 4.3.1.1 Add analysis of AEs of special | Summarize common AEs associated |
| | | Section 4.3.1.2: Add 'and a Toeplitz covariance structure' to the SAS PROC MIXED details | with ARI treatment Align with protocol v2.0 |


## ARAMON V3.0

| <b>_</b> | 1 | | <u></u> |
|---|---|---|---|
| | | Section 4.5: Remove language related to | Laboratory measures are not graded in |
| | | grading of laboratory measures | this study |
| | | Section 4.5.2 Remove TEAEs with incidence of | Not meaningful with the sample size of |
| | | at least 5% table | the study |
| | | Section 4.5.2 Add drug related TEAEs; add a | Elaborate safety findings |
| | | comprehensive list of safety tables planned | |
| | | Section 4.6.1: Add free testosterone as | Explore the treatment effect of |
| | | exploratory analysis for lead-in phase primary | darolutamide on free testosterone |
| | | analysis | |
| | | Section 4.6.1: Remove FACT-P and exploratory | Prioritizing the important endpoints for |
| | | endpoints from lead-in primary analysis | decision making to go into the |
| | | | randomized phase |
| | | Section 6.1.1: Add Discontinued from treatment | Align with clarification on active follow- |
| | | along with the primary reason for discontinuation | up in protocol v2.0 |
| | | in place of participants continued after treatment | |
| | | discontinuation | |
| | | Section 6.1.2: Revise age groups | Align with ICH E7 Q&A (2010) |
| | | | recommendations |
| | | Section 6.1.2: Add time from first progression | Assess the disease progression |
| | | and most recent relapse to first dose | |
| | | Section 6.1.2: Add eGFR | Assess renal function |
| | | Section 6.1.2: Revise list of baseline lab | Align with the endpoints planned to |
| | | variables | assess and to prioritize the important |
| | | | endpoints for lead-in primary analysis |
| | | Appendix 5: Add PROC for primary endpoint | Clarification and corrections |
| | | analysis and corrections to the current code | |
| | | Appendix 6: Corrections to the current code | Corrections |
| 3.0 | 06 MAR 2024 | Section 4.5.2: Add Treatment-emergent study | Assess the worst grades of each |
| | | drug-related adverse events of feminizing side | feminizing side-effect |
| | | effects by MedDRA SOC and PT and worst | |
| | | CTCAE grade | |
| | | Section 4.6.1: Add PSA analysis with non- | Since the study is ongoing |
| | | confirmed responses for Lead-in primary | |
| | | analysis | |
| | | Section 4.6.1: Add median treatment duration for | Study how long subjects were on |
| | | Lead-in primary analysis | treatment at the time of analysis |
| | | Section 4.6.2: Add Feminizing side effects | Assess the adverse events profiles for |
| | | analysis by <=50% and >50% week 12 | subgroups |
| | | testosterone increase subgroups | |
| | | Section 6.1.2: Remove baseline value | The important baseline summaries |
| | | presentation for Sex hormones and Fat and | needed for decision making are in their |
| | | glucose metabolism for lead-in primary analysis | respective endpoint tables |
| | | Change AEs of special interest to AEs of special | For consistency across darolutamide |
| | | topics | studies |

ARAMON V3.0 

#### 1. Introduction

The SAP describes the planned analyses of the ARAMON study, a Phase 2, Randomized, Open-label study of Darolutamide or Enzalutamide Monotherapy on Testosterone Levels in Men with Hormone-Naïve Prostate Cancer. Details included in the SAP include a description of endpoints, a brief description of the study design, analysis sets and statistical methodology.

ARAMON is designed to evaluate the efficacy and safety of treatment of men with hormone sensitive prostate cancer experiencing biochemical recurrence (BCR) with darolutamide or enzalutamide monotherapy. Efficacy outcomes measured will include serum testosterone levels, PSA levels and hormonal changes derived from the androgen axis including endocrine and energy metabolism markers and changes in bone mineral density. Study will also evaluate safety and quality of life, as well as fitness and physical function.

The analysis of the study will be conducted at three data cuts expected after about 12 weeks after start of darolutamide therapy for the lead-in phase, after 12 weeks post-randomization in the randomized phase and at end of the randomized phase. Table, figure and listing specifications are contained in a separate document.

Currently, there are no changes to the analyses described in the protocol amendment 1.0.

ARAMON V3.0 

# 1.1. Objectives, Endpoints, and Estimands

Table 1-1: Lead-in phase objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the impact of darolutamide | Change in serum testosterone level from |
| on serum testosterone level | baseline to week 12 |
| over a 12-week intervention period | |
| Secondary | |
| To evaluate the impact of darolutamide | Change in serum testosterone level from |
| monotherapy on serum testosterone level over | baseline at week 24 and 52 |
| the course of a 52-week intervention period | |
| Assess PSA response rate | Serum PSA Week 4, 12, 24, 36, 52 |
| To assess safety of darolutamide monotherapy | AE assessments using NCI CTCAE (v.5.0) |
| in participants with hormone-naïve prostate | |
| Cancer with BCR | |

Abbreviations: BCR-Biochemical Recurrence, NCI CTCAE-National Cancer Institute Common Terminology Criteria for Adverse Events, PSA Prostate Specific Antigen.

Table 1-2: Randomized Phase Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To compare the effects of treatment with darolutamide vs. enzalutamide monotherapy on serum testosterone level over a 12-week intervention period | Change in serum testosterone level from baseline to week 12 |
| Secondary | |
| To compare the effect of darolutamide vs. enzalutamide monotherapy on serum testosterone level over the course of a 52-week intervention period | Change in serum testosterone level from baseline at week 24 and 52 |
| Measure changes in markers of endocrine function related to sex hormones | Changes in the blood levels of sex hormones (DHT, DHEA, SHBG, LH, FSH, Androstenedione, Prolactin, Estradiol) |
| Measure changes in markers of components of fat and glucose metabolism | Changes blood levels of Total cholesterol, High-<br>density and low-density lipoproteins,<br>Triglycerides, Haemoglobin A1C, Fasting insulin,<br>Fasting glucose, Fat body mass, Lean body mass |
| Assess PSA response rate | Serum PSA Week 4, 12, 24, 36, 52 |
| To assess safety and QOL of darolutamide vs. enzalutamide monotherapy in participants with hormone-naïve prostate Cancer with BCR | AE assessments using NCI CTCAE (v.5.0) and FACT-P |
| Exploratory | |
| Evaluate changes in Bone turnover | Markers of bone turnover:<br>BSAP, CTX, DEXA scan |
| Physical function* | Subjective physical function: Godin – 4 questions, PROMIS Fatigue – 8 questions, PROMIS Physical – 6 questions, Self- Efficacy – 9 questions |

Abbreviations: A1C-glycated (hemoglobin), AE adverse events, BCR-Biochemical Recurrence, BSAP bone specific alkaline phosphatase, CTX C-telopeptid, DHEA-dehydroepiandrosterone, DHT-dihydrotestosterone, DEXA dual energy x-ray absorptiometry, FACT-P Functional Assessment of Cancer Therapy – Prostate Cancer, FSH-follicle-stimulating hormone, LH-luteinizing hormone, NCI CTCAE-National Cancer Institute-Common Terminology Criteria for Adverse Events, PSA-Prostate-specific antigen, QOL Quality of life, SHBG- sex hormone-binding globulin, PROMIS Patient-Reported Outcomes Measurement Information System.\*The physical function assessments might be modified.

ARAMON V3.0 

# 1.2. Study Design

## 1.2.1 Overall Design

This is a two-stage open-label phase 2 study with a lead-in single-arm phase and the randomized phase, to assess the impact of androgen receptor inhibitor (ARI) darolutamide or enzalutamide as a monotherapy treatment on serum testosterone levels in men with hormone-naïve prostate cancer experiencing BCR. The study design is shown in Figure 1-1.

Figure 1-1: Overall Design



Abbreviations: ECOG Eastern cooperative oncology group, PC prostate cancer, PSADT PSA doubling time.

In the lead-in phase, participants will be treated with darolutamide (600 mg twice daily). The primary analysis of the lead-in phase will occur when the last participant in the lead-in phase has been on treatment for 12 weeks, unless the participant discontinued due to lost to follow-up, withdrawal, or death. Analysis will be based on a date-based data cut in which the cutoff date will be the last participant week 12 visit date.

The study team will review the findings from the lead-in phase and provide input on interpretation of the results from the lead-in phase. This will help guide a decision on go/no-go with the randomized phase as well as potential changes in the study design for the randomized phase by the sponsor.

In case of the decision to proceed in the randomized phase, participants will be randomized in a 1:1 ratio to receive either darolutamide (600 mg twice daily) or enzalutamide (160 mg once daily). The primary analysis of randomized phase will be conducted when the last participant in the randomized phase has been on treatment for at least 12 weeks. Similar to lead-in phase the analysis will be based on a date-based data cut.

The final analysis for both phases of the study will occur when last participant in the randomized phase has been on treatment for at least 52 weeks, unless the participant discontinued due to lost to follow-up, withdrawal, or death.

The overall sample size across the two phases is expected to be about 65 participants.

The study will comprise the following consecutive periods: Screening, Treatment, and Active Follow–up.

ARAMON V3.0 

## 1.2.1.1 Screening period

After the participant has signed the Informed Consent Form (ICF), the screening period will begin from the date of signed ICF to up to 28 days before start of study intervention (date of first dose). Enrolled participants include those who signed the informed consent form, met all inclusion and none of the exclusion criteria, and are eligible for the first dose of study drug. The IWRS system will assign a unique participant ID to an enrolled participant.

#### 1.2.1.2 Treatment period

The treatment period is defined as the time from the administration of first dose of study treatment until 52 weeks or unacceptable toxicity, withdrawal of consent, investigator's decision to stop therapy for the participant, participant decision to stop therapy, sponsor's decision to terminate the study, or death.

End of treatment (EOT) visit takes place 30 days (+7 days) after the last dose.

#### 1.2.1.3 Active Follow-up period

When the participant's treatment is discontinued before completing week 52 treatment, the participant will continue assessments until week 52. This follow-up period is defined as the Active Follow-up period.

## 1.2.2 Participant completion of study

A participant is considered to have completed the study if he has completed all periods of the study (see protocol Table 1.3 for lead-in phase, Table 1.4 for randomized phase, and Table 1.5 for active follow-up period), unless the participant discontinued due to lost to follow-up, withdrawal, or death.

#### 1.2.3 End of Study Definition

The end of the study is defined as the date of the LPLV in the study.

LPLV of the study is reached when all participants have completed the last scheduled procedure shown in the Schedule of Activities including the active follow-up period.

ARAMON V3.0 

# 2. Statistical Hypotheses

The core questions to be addressed in the two phases of the study are described in the following sections.

## **Lead-in Phase**

Descriptive analyses will be provided for the lead-in phase without formal hypothesis testing.

## **Randomized Phase**

The randomized phase will test the Null Hypothesis of no difference between the Darolutamide arm and the Enzalutamide arm on the primary endpoint of mean percent change in Testosterone from baseline to week 12, against the alternative hypothesis of a difference between arms at a two-sided 0.05 level. For mean percent changes of  $\Delta_D$  and  $\Delta_E$  in the Darolutamide and Enzalutamide arms these hypotheses can be expressed as

$$H_0$$
:  $\Delta_D = \Delta_E \text{ vs. } H_1$ :  $\Delta_D \neq \Delta_E$ 

# 2.1. Multiplicity Adjustment

Not applicable as there are no co-primary endpoints or interim analyses requiring special means for the control of the overall false positive error rate.

ARAMON V3.0 

# 3. Analysis Sets

For purposes of analysis, the following populations are defined:

Table 3-1: Populations for analyses: Lead-in phase

| Population | Description |
|---|---|
| Screened | All participants who sign the informed consent form |
| Evaluable | All enrolled participants having testosterone data at baseline and Week 12. Enrolled participants include those who signed informed consent and met all inclusion and none of the exclusion criteria. |
| Safety | All enrolled participants who received any darolutamide post-enrollment regardless of their eligibility for the study. |

Table 3-2: Populations for analyses: Randomized Phase

| Population | Description |
|---|---|
| Screened | All participants who sign the informed consent form |
| Evaluable | All randomized participants having testosterone data at baseline and week 12 who signed informed consent and met all inclusion and none of the exclusion criteria. |
| Safety | All randomized participants who received any quantity of study intervention, regardless of their eligibility for the study. The safety evaluation will be performed based on the intervention actually received. |

Final decisions regarding the assignment of participants to analysis sets will be made during the review of study data and documented in the final list of important deviations, validity findings and assignment to analysis set(s).

ARAMON V3.0 

# 4. Statistical Analyses

## 4.1. General Considerations

All baseline variables will be reported using the appropriate statistics: categorical variables by frequency tables (frequencies and percentages) and continuous variables by sample statistics (i.e., mean, standard deviation, minimum, median, quartiles, and maximum). The number of participants screened will be summarized for both the lead-in and randomized cohorts.

The efficacy related endpoints will be evaluated in the evaluable population while the safety endpoints will be evaluated in the safety population.

Efficacy endpoints will consider data until last dose of study drug (while on treatment).

#### 4.1.1 Analysis junctures

The analyses for this study will occur at three junctures as described in section 1.2.1. The endpoints analyzed at each juncture will be as follows:

- For primary analysis of the lead-in phase: Primary endpoint of percent change in testosterone; PSA responses at 4 and 12 weeks; incidence of treatment emergent adverse events with emphasis on feminizing side effects.
- For primary analysis of the randomized phase: Primary endpoint of percent change in testosterone; PSA responses at 4 and 12 weeks; other sex hormone changes at 4 and 12 weeks; components of fat and glucose metabolism at 4 and 12 weeks; incidence of treatment emergent adverse events with emphasis on feminizing side effects.
- Final analysis: Separate analyses will be performed for the lead-in phase and the randomized phase of the study. For the lead-in phase, summaries for visits after 12 weeks will be presented for testosterone, PSA, and safety endpoints. For the randomized phase, summaries at the visits after week 12 will be presented for testosterone, sex hormones, components of fat and glucose metabolism, and additional efficacy and safety endpoints.

#### 4.1.2 Handling missing data

All missing or partial data will be presented in the participant data listing as they are recorded on the Case Report Form. Except as noted, missing data will not be estimated or carried forward in any statistical analysis.

When appropriate, the following rules will be implemented so as not to exclude participants from statistical analyses due to missing or incomplete data:

## <u>Incomplete death dates:</u>

Every effort should be made to resolve incomplete or missing dates during the course of the study (i.e., edit checks, data cleaning/monitoring etc.). However, in rare circumstances, missing parts of either the censoring date or the event date may occur where an imputation algorithm must be defined. In general, the following rule should be followed: A missing month or year is not acceptable. To impute a value for day, day 15 of the month will be used for the calculation.

ARAMON V3.0 

#### Partial or missing AE dates:

Refer to Appendix 1: Imputation rule for partial missing dates for the imputation rule for incomplete AE dates.

## **Laboratory Assessments:**

To facilitate the transformation of the data, the least detectable values of Testosterone and other laboratory values will be used when the baseline data notes a less than detectable value. When such a value is not uniformly available across sites, then the lowest value of the laboratory analyte across participants at baseline in the data cut will be used.

#### FACT-P Questionnaire:

For FACT-P, total scores and subscale scores (physical well-being, social/family well-being emotional well-being, and functional well-being) will be assessed. Where there are missing items, subscale scores will be prorated if >50% of items on subscale are completed. This will be done by multiplying the sum of the subscale by the number of items in the subscale, then dividing it by the number of items answered. If  $\leq$ 50% of the items are answered for any domain, then the score of that domain will be set to missing (see scoring of FACT-P in Appendix 2: Scoring procedures for FACT-P). The total score will be set to missing if the related overall item response rate is less than or equal to 80% (without prorated subscale items). In addition, a total score will only be calculated if all the component subscales have valid scores.

The statistical evaluation will be performed by using the software SAS (release 9.4 or higher; SAS Institute Inc., Cary, NC, USA. All data will be presented in the participant data listing as they are recorded on the Case Report Form (CRF), i.e., partially missing data will appear as such.

#### 4.1.3 Data rules

In case of repeated measurements over multiple dates per time point,

- For baseline, the nearest visit (scheduled or unscheduled) to the start of the study drug administration will be used;
- For post-baseline measures, the scheduled visit will be used. Unscheduled visits will be used if there are no scheduled visits then the first unscheduled visit will be used.

If there are repeated measurements per time point on the same day (e.g., laboratory values, vital signs, etc.),

- For baseline, the latest measurement will be used;
- at any post baseline time point, the first measurement at the visit will be used.

# 4.2. Primary Endpoint Analysis

The primary endpoint, percent change in testosterone, is defined in Section 1.1. The primary endpoint for both phases will be analyzed using a natural logarithm transformation consistent with sample size assessments in Section 5 given a distribution for the endpoint which is skewed right. Further, the percent change endpoint is a re-scaled fold change from baseline statistic for which such a transformation is often conducted. The mean fold change and

ARAMON V3.0 

percent change estimates are interpretable as geometric means given the logarithmic transformation.

The primary endpoint will be analyzed in the evaluable population.

#### 4.2.1 Main Analytical Approach

The primary endpoint for the lead-in phase will be analyzed at 12 weeks after start of darolutamide for the last participant in the lead-in phase. If the study continues into the randomized phase, the primary endpoint analysis for the randomized phase will be conducted 12 weeks after start of study treatment for the last participant in the randomized phase.

#### 4.2.1.1 Lead-in Phase

The participant testosterone levels at baseline and week 12 will be transformed to natural logarithm values. The mean and 95% Confidence Interval of the differences between the week 12 and baseline values will be computed and back transformed by exponentiation to obtain the mean fold change  $M_F$  with its 95% Confidence Interval [ $L_F$ ,  $U_F$ ]. The mean percent change  $\Delta$  can be obtained as  $\Delta = 100*(M_F-1)$  with Confidence Interval [ $100*(L_F-1)$ ,  $100*(U_F-1)$ ]. In addition to the estimated mean percent change and its confidence interval, summary statistics will include the mean fold change with confidence intervals, and the mean, standard deviation, median, quartiles, minimum, and maximum of percent change computed from the raw week 12 and baseline testosterone values.

#### 4.2.1.2 Randomized Phase

The participant level differences between the natural log transformed testosterone values at week 12 and baseline will be computed. These differences will be compared across the darolutamide and enzalutamide arms using a two-sample t-test. SAS code will be similar to code shown in Appendix 4: Randomized phase primary endpoint analysis for natural logarithm transformed Testosterone. Two-sided p-values from this t-test will be reported to assess whether the null hypothesis can be rejected in favor of the alternate hypothesis described in Section 2. Additionally, the estimated difference between darolutamide and enzalutamide and the 95% confidence limits from the t-test will be back transformed by exponentiation to obtain the ratio of the fold change in testosterone values from baseline for darolutamide to that for enzalutamide and the confidence limits for this estimate. Within treatment group, mean percent change and confidence intervals as well as other summary statistics described for the lead-in phase will also be reported.

# 4.3. Secondary Endpoint Analysis

All secondary endpoints, as described in Section 1.1, will be analyzed in the evaluable population except for the safety endpoints, which will be analyzed in the safety population.

#### 4.3.1 Main Analytical Approach

The secondary endpoints summarized at each juncture of the study are detailed in Section 4.1. The analysis approach for each secondary endpoint at each phase is as follows.

#### 4.3.1.1 Lead-in Phase

• Testosterone at weeks 24 and 52:

ARAMON V3.0 

The differences between the log transformed data at the visit and baseline will be estimated with 95% Confidence Intervals using SAS PROC MIXED with the ESTIMATE statement. These will be transformed to mean percent change and 95% confidence intervals using the same steps as for the primary analysis in the lead-in phase. SAS code will be similar to code shown in Appendix 5: Lead-in phase analysis for natural logarithm transformed Testosterone and other endpoints using the log transformation. Results for testosterone at week 24 and 52 will be summarized in a similar manner to the primary endpoint and depicted graphically over time with 95% confidence intervals at each visit.

#### • PSA responses:

## o Undetectable PSA response

Undetectable PSA is defined as a baseline PSA value above the 0.2 ng/mL detection limit and a post baseline PSA level below 0.2 ng/mL, confirmed by a second subsequent PSA value below 0.2 ng/mL 3 or more weeks later, with all potential PSA values between the initial date and the confirmation date below 0.2 ng/mL.

The undetectable PSA response is defined as the number of participants with undetectable PSA divided by the total number of participants evaluable. The undetectable PSA response will be summarized at 4, 12, 24, 36 and 52 weeks.

#### o PSA50, PSA90

PSA50 is defined as a baseline PSA value above the 0.2 ng/mL detection limit and a post baseline  $\geq$ 50% reduction of the PSA level compared to the baseline value, confirmed by a second subsequent PSA value with a  $\geq$ 50% reduction from baseline 3 or more weeks later, with all potential PSA values between the initial date and the confirmation date showing a  $\geq$ 50% reduction from baseline. PSA90 is defined in the same way with 90% reduction.

The PSA50 response is defined as the number of participants with PSA50 divided by the total number of participants evaluable. The PSA90 response is defined the same way. PSA50 and PSA90 will be summarized at 4, 12, 24, 36 and 52 weeks.

In addition, descriptive statistics will be provided for PSA maximum percent decline of  $\geq$  50%,  $\geq$  90% from baseline at any time on study.

#### • Analysis of AEs:

All grades of the feminizing side effects of gynecomastia (including breast enlargement, breast mass, breast swelling), breast tenderness/pain, nipple pain, and hot flush will be summarized using frequencies and percentages. Incidence of AEs of special topics (Bone fractures excluding pathological fractures, Cerebral ischemia, Diabetes mellitus and Hyperglycaemia, Fall, Fatigue/ asthenic conditions, Weight decreased, Rash, Seizure, Hypertension, Vasodilatation and flushing, Mental impairment disorders, Depressed mood disorders, Breast disorders/gynecomastia, Cardiac disorders, Cerebral and intracranial hemorrhage) associated with ARI treatment will also be presented.

#### 4.3.1.2 Randomized Phase

#### • Testosterone at weeks 24 and 52:

The differences between the log transformed data at the visit and baseline will be compared across treatment groups with 95% Confidence Intervals using SAS PROC MIXED with the SLICE option and a Toeplitz covariance structure. These will be

ARAMON V3.0 

transformed to the ratio of the fold change from baseline for darolutamide to that for enzalutamide and 95% confidence intervals using the same steps as for the primary analysis in the randomized phase. SAS code will be similar to code shown in Appendix 6: Randomized phase analysis for natural logarithm transformed Testosterone and other endpoints using the log transformation. Results will be summarized in a similar manner to the primary endpoint and will be summarized graphically using the mean percent change over time with 95% confidence intervals at each visit by treatment group, flagging visits where differences are significant at the nominal 0.05 and 0.01 levels.

#### • Sex hormones:

Will be analyzed at week 4, 12, 24 and 52 similar to testosterone.

#### • Components of fat and glucose metabolism:

Will be analyzed at week 4, 12, 24 and 52 similar to testosterone.

#### PSA responses

Will be compared descriptively across treatments at weeks 4, 12, 24, 36 and 52 using frequencies and percentages.

#### • FACT-P

Differences in the FACT-P prostate cancer subscale and total will be summarized at each visit using PROC Mixed with the SLICE option, and the mean subscale and total scores will be depicted graphically over time with 95% confidence intervals at each visit by treatment group, flagging visits where differences are significant at the nominal 0.05 and 0.01 levels. The scoring procedure for FACT-P is elaborated in Appendix 2: Scoring procedures for FACT-P.

#### • Analysis of AEs:

All grades of the feminizing side effects of gynecomastia (including breast enlargement, breast mass, breast swelling), breast tenderness/pain, nipple pain, and hot flush, will be summarized using frequencies and percentages by treatment group.

# 4.4. Other Exploratory Endpoints

#### • Markers of bone turnover:

Will be analyzed for the randomized phase as described for the sex hormones and components of fat and glucose metabolism in Section 4.3.1.2.

#### • Physical function measures:

Will be summarized graphically as described for the FACT-P subscale in Section 4.3.1.2. The scoring procedures for PROMIS physical function questionnaires are elaborated in Appendix 3: Scoring for PROMIS.

# 4.5. Safety Analyses

All safety analyses will be descriptive and will be performed on the safety population. Safety data will be summarized descriptively for the lead-in phase and by treatment group for the randomized phase.


All AEs will be coded using the latest version prior to database lock of the Medical Dictionary for Regulatory Activities (MedDRA).

NOTE: AEs will be presented with their worst NCI-CTCAE grade.

#### 4.5.1 Extent of Exposure

Study drug is defined as darolutamide for the lead-in, and darolutamide and enzalutamide for the randomized phase. As a rule, trailing "0 mg" records, which are not followed by any positive amount of drug, will not be included in the calculation of any drug duration or amount. Similarly, trailing "drug interruptions" will not be used in statistical tables. Interruption becoming permanent study treatment discontinuation is not accounted as an interruption.

Descriptive statistical summaries will be provided for the for the following variables:

• Overall time under treatment (or treatment duration)

Including time off drug and dose interruptions. It will be calculated in days and presented in months as (date of the last dose of any study treatment – date of the first dose of any study treatment + 1) / 30.44.

Actual dose per day

Actual dose per day = total amount of dose / number of days with intake > 0

• Total amount of dose

Total amount of dose = sum of dose received over total time under treatment

• Percent of planned dose received.

Percent of planned dose received = total amount of dose [mg] / planned dose [mg] \* 100%; planned dose is sum of the intended initial dose according to protocol over total time under treatment.

#### 4.5.2 Adverse Events

Treatment-emergent AE (TEAE) is defined as any event arising or worsening after the first dose of study drug until 30 days after the last dose of study drug.

An overview of TEAEs will be summarized for the appropriate safety analysis set at the three data cuts. The following summaries will be done.

- Overview of TEAEs
- TEAEs by MedDRA ad worst CTCAE grade
- TEAEs by MedDRA ad worst CTCAE grade 3, 4 or 5
- TEAEs: number of subjects by primary SOC and PT
- TEAEs leading to permanent discontinuation of study drug: number of subjects by primary SOC and PT
- Number of subjects with TEAE by PT in decreasing order
- Drug-related TEAEs: number of subjects by primary SOC and PT

• Drug-related TEAEs leading to permanent discontinuation of study drug: number of subjects by primary SOC and PT


- Number of subjects with drug-related TEAE by PT in decreasing order
- SAEs: number of subjects by primary SOC and PT
- TESAEs: number of subjects by primary SOC and PT
- Drug-related TESAEs: number of subjects by primary SOC and PT
- TE non-SAEs (excluding TESAEs): number of subjects by primary SOC and PT

Additionally, feminizing side effects as described in Section 4.3, will be summarized by

- Overview of TEAEs of feminizing side effects
- Number of subjects with TEAEs of feminizing side effects by PT in decreasing order
- Treatment-emergent study drug-related adverse events of feminizing side effects by MedDRA SOC and PT and worst CTCAE grade
- Number of subjects with TEAEs of feminizing side effects leading to permanent discontinuation of study drug by PT in decreasing order
- Number of subjects with drug-related TEAEs of feminizing side effects by PT in decreasing order
- Number of subjects with drug-related TEAEs of feminizing side effects leading to permanent discontinuation of study drug by PT in decreasing order
- SAEs of feminizing side effects: number of subjects by primary SOC and PT
- TESAEs of feminizing side effects: number of subjects by primary SOC and PT
- Drug-related TESAEs of feminizing side effects: number of subjects by primary SOC and PT

AEs of special topics will be summarized by

• Number of subjects with special topics for adverse events

## 4.6. Other Analyses

#### 4.6.1 Lead-in Phase Analyses

For the lead-in phase primary analysis: change in free testosterone from baseline to week 12, will be analyzed similar to serum testosterone. PSA response analysis summarized in section 4.3.1.1 will be repeated with non-confirmed PSA responses. Data collected on the CRF for Serum and Free testosterone, PSA, sex hormones, fat and glucose metabolism will be summarized in spider plots to support any changes to data collection for the randomized phase, or for additional support of the randomized phase findings. The median treatment duration will be presented in months. For subjects ended treatment before the data cut-off date, duration will be 'last dose date – first dose day +1'. For subjects on treatment by the day of data cut-off, the duration will be 'data cutoff date – first dose day +1'.

For the lead-in phase final analysis: for the sex hormones and the components of fat and glucose metabolism at weeks 4, 12, 24 and 52, the differences between the log transformed

ARAMON V3.0 

data at the visit and baseline will be estimated with 95% Confidence Intervals using SAS PROC MIXED with the ESTIMATE statement. These will be transformed to mean percent change and 95% confidence intervals using the same steps as for the primary analysis in the lead-in phase. SAS code will be similar to that shown in Appendix 5: Lead-in phase analysis for natural logarithm transformed Testosterone and other endpoints using the log transformation. Sex hormones and fat and glucose metabolism endpoints will be depicted graphically over time with 95% confidence intervals at each visit.

The FACT-P prostate cancer subscale scores will be summarized at each visit using PROC Mixed with the ESTIMATE statement and depicted graphically over time with 95% confidence intervals at each visit.

The physical function scores will be summarized graphically using the methods described above for FACT-P.

#### 4.6.2 Subgroup Analyses

For lead-in phase primary analysis:

Overview of treatment-emergent adverse events of feminizing side effects, Number of subjects with treatment-emergent study drug-related adverse events of feminizing side effects by preferred term in decreasing order, Number of subjects with treatment-emergent study drug-related adverse events of feminizing side effects by worst CTCAE grade will be presented for the <=50% and >50% week 12 testosterone increase subgroups.

# 4.7. Interim Analyses

No group sequential interim analyses are planned. However, the analysis will be conducted at three junctures as described in Section 1.

# 4.8. Changes to Protocol-planned Analyses

There are no changes to the analyses described in the protocol.

ARAMON V3.0 

# 5. Sample Size Determination

The sample sizes corresponding to the planned analysis methodology are provided below.

#### Lead-in Phase

Approximately 25 participants will be assigned to darolutamide to achieve at least 20 evaluable participants. This sample size will help estimate the mean percent change in serum testosterone level at 12 weeks with a 95% confidence interval having a half-width of no more than 25%, assuming a true mean percent increase of less than 45% and a standard deviation of 65%. This assessment uses a log normal distribution for percent change.

## **Randomized Phase**

Contingent on the results of the evaluation in Section 1.2.1, the randomized phase statistical assumptions may be revised, or the study could be terminated after lead-in.

Should the study continue to the Randomized phase unmodified, a maximum of 40 participants (20 per arm) will be randomly assigned to study treatment (darolutamide or enzalutamide) such that approximately 34 evaluable participants complete the study. The randomized stage will require a sample size of 20 per group to provide 85% power to test the null hypothesis of no difference between groups on mean percent change at the two-sided 0.05 level. This assessment is based on a mean percent change in Testosterone from baseline and Standard Deviation for the Darolutamide arm of 45% and 65% versus 110% and 75% respectively for Enzalutamide and assumes a log normal distribution for percent change.

ARAMON V3.0 

# 6. Supporting Documentation

# **6.1.** Population Characteristics

# 6.1.1 Disposition of participants

Overall summaries will be presented for the lead-in phase, and by treatment arm as well for the randomized phase.

The number and the percentages of participants for the following will be summarized:

- Screened, Evaluable and Safety populations
- Discontinued from screening along with the primary reason for discontinuation
- Discontinued from treatment along with the primary reason for discontinuation
- Discontinued from active follow-up along with the primary reason for discontinuation

## 6.1.2 Demographics and baseline characteristics

Overall descriptive summaries of demographics and baseline characteristics will be presented for the lead-in phase, and by treatment arm as well for the randomized phase on the Evaluable population.

The following demographic data will be summarized:

- Age (years)
- Age category ( $<65, 65-74, 75-84, \ge 85 \text{ years}$ )
- Ethnicity
- Race
- Weight (kg)
- BMI (kg/m<sup>2</sup>)

The following baseline characteristics will be summarized:

- ECOG Performance Status
- Stage of prostate cancer at initial diagnosis
- Gleason score of prostate cancer (<8,  $\ge$ 8) at initial diagnosis
- Stage of prostate cancer at study entry
- Serum testosterone group ( $< 150 \text{ ng/dL}, \ge 150 \text{ ng/dL}$ )
- Time from initial diagnosis to first dose of study drug (months)
- Bone lesions at baseline (Y/N)
- Number of bone lesions at baseline
- Hepatic function at baseline:
  - o Normal: Total bilirubin and AST  $\leq$  upper limit of normal (ULN)

ARAMON V3.0

o Mild impairment: Total bilirubin > ULN to 1.5 x ULN or (Total bilirubin ≤ ULN and AST > ULN)


- o Moderate impairment: Total bilirubin > 1.5 to 3 x ULN, any AST
- Severe impairment: Total bilirubin > 3 x ULN, any AST.
- Estimated glomerular filtration rate (eGFR) at baseline:
  - o eGFR =  $[(140 Age) \times Weight/(72 \times Creatinine)]$ .

The following baseline lab values, assessed in secondary and exploratory endpoints, will be summarized in a separate baseline table:

- Serum testosterone
- Free testosterone
- PSA
- Sex hormones
- Fat and glucose metabolism
- FACT-P
- Bone turnover
- Physical function

## 6.1.3 Prior anti-cancer therapies

The prior systemic anti-cancer therapy summaries and summaries of prior radiotherapies and surgeries will be presented for the lead-in phase, and by treatment arm as well for the randomized phase on the Evaluable population.

#### 6.1.4 Important protocol deviations

The number of participants with important protocol deviations will be presented by treatment arm and overall. The frequencies of each important protocol deviation will be presented by treatment arm and overall. All COVID-19 pandemic related protocol deviations are considered important protocol deviations and will be presented by treatment arm and overall.


ARAMON V3.0

# **Appendix 1: Imputation rule for partial missing dates**

| Partial Dates<br>Imputation<br>Rule | Impute partial AE Start Date | Impute partial AE Stop Date |
|---|---|---|
| The day missing only | IF AESTDT year and month is same as TRTSDT year and month, then impute AESTDT= TRTSDT | IF AEENDT year and month is same as last known alive date (LKAD) year and month, then impute AEENDT= LKAD |
| | ELSE IF AESTDT year and month is before TRTSDT year and month, then AESTDT= last date of the month | ELSE impute AEENDT= last date of the month |
| | ELSE IF AESTDT year and month is after TRTSDT year and month, then AESTDT= first date of the month | |
| Both day and month missing | IF AESTDT year is same as TRTSDT year, then impute AESTDT=TRTSDT | IF AEENDT year is same as last known alive date (LKAD) year, then impute AEENDT= LKAD |
| | ELSE IF AESTDT year is before TRTSDT year, then impute AESTDT=31DECYYYY | ELSE impute AEENDT=31DECYYYY |
| | ELSE IF AESTDT year is after TRTSDT year, then impute AESTDT=01JANYYYY | |
| Completely missing | No need to impute, try to query the sites by DM | No need to impute, try to query the sites by DM |
| Additional criteria to meet | <ol> <li>AE start date &lt;= AE stop date</li> <li>The imputed dates &lt;= last known alive date (LKAD)</li> <li>If TRTSDT is missing, use RANDDT as reference date</li> </ol> | |

# **Appendix 2: Scoring procedures for FACT-P**

# **FACT-P Scoring Guidelines** (Version 4)

Instructions: 1. F

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated and sum individual items to obtain a score.

ARAMON V3.0

3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.


- 4. Add subscale scores to derive total scores (TOI, FACT-G & FACT-P).
- 5. The higher the score, the better the QOL.

| <b>Subscale</b> | <b>Item Code</b> | Revers | e item? | <u>Item response</u> | Item Sc | <u>ore</u> |
|---|---|---|---|---|---|---|
| PHYSICAL | GP1 | 4 | _ | | = | |
| WELL-BEING | GP2 | 4 | _ | | = | |
| (PWB) | GP3 | 4 | _ | | = | |
| (2 11 2) | GP4 | 4 | _ | | = | |
| | GP5 | 4 | _ | | = | |
| Score range: 0-28 | GP6 | 4 | _ | | = | |
| | GP7 | 4 | _ | | = | |
| | | • | | | | |
| | | | | Sum individual item | scores: | |
| | | | | Multip<br>e by number of items an | oly by 7: | |
| | | | Divid | e by number of items an | iswered: | =PWB subscale |
| <u>score</u> | | | | | | |
| SOCIAL/FAMILY | GS1 | 0 | + | | = | |
| WELL-BEING | GS2 | 0 | + | | = | |
| (SWB) | GS3 | 0 | + | | = | |
| (2.77) | GS4 | 0 | + | | = | |
| | GS5 | 0 | + | | = | |
| Score range: 0-28 | GS6 | 0 | + | | = | |
| Score range. 0 20 | GS7 | 0 | + | | = | |
| | | | | | | <del></del> |
| | | | | Sum individual item | scores: | |
| | | | | Multip | ly by 7: | |
| | | | Divide | by number of items an | swered: | =SWB subscale |
| <u>score</u> | | | | | | |
| <b>EMOTIONAL</b> | GE1 | 4 | - | | = | |
| WELL-BEING | GE2 | 0 | + | | = | |
| (EWB) | GE3 | 4 | - | | = | |
| | GE4 | 4 | - | | = | |
| Score range: 0-24 | GE5 | 4 | - | | = | |
| Score range. 0-24 | | | | | | |
| | GE6 | 4 | - | | = | |
| | | | | Sum individual item | scores: | |
| | | | | Multip | ly by 6: | |
| | | | Divide | by number of items an | swered: | = <u>EWB subscale</u> |
| <u>score</u> | | | | | | |
| FUNCTIONAL | GF1 | 0 | + | | =_ | |
| WELL-BEING | GF2 | 0 | + | | = | |
| (FWB) | GF3 | 0 | + | | = | |
| | GF4 | 0 | + | | = | |
| | GF5 | 0 | + | | = | |
| Score range: 0-28 | GF6 | 0 | + | | = | |
| | GF7 | 0 | + | | = | |
| | | | | Sum individual item | scores: | |

ARAMON V3.0 

| Multiply by 7: | |
|-------------------------------------|---------------------|
| Divide by number of items answered: | =FWB subscale score |

| <b>Subscale</b> | <b>Item Code</b> | Reverse ite | <u>m?</u> | <u>Item response</u> | <b>Item Score</b> |
|---|---|---|---|---|---|
| PROSTATE | C2 | 4 | _ | | = |
| CANCER | C6 | 0 | + | | = |
| SUBSCALE | P1 | 4 | - | <del></del> | = |
| (PCS) | P2 | 4 | - | | = |
| | P3 | 4 | - | | = |
| 0.40 | P4 | 0 | + | | = |
| Score range: 0-48 | P5 | 0 | + | | = |
| | P6 | 4 | - | | = |
| | P7 | 4 | - | | = |
| | BL2 | 4 | - | | = |
| | P8 | 4 | - | | = |
| | BL5 | 0 | + | | = |

Sum individual item scores:\_\_\_\_\_ Multiply by 12: \_\_\_\_\_ Divide by number of items answered: \_\_\_\_\_=PC Subscale score

#### To derive a FACT-P Trial Outcome Index (TOI):

Score range: 0-104  $\frac{+}{(PWB \text{ score})} + \frac{+}{(FWB \text{ score})} + \frac{-}{(PCS \text{ score})} = \frac{-}{-} = \frac{-}{FACT-P \text{ TOI}}$ 

#### To Derive a FACT-G total score:

Score range: 0-108

+ \_\_\_\_ + \_\_\_ + \_\_\_ + \_\_\_ = \_\_\_ = FACT-G Total score

(PWB score) (SWB score) (EWB score)

#### To Derive a FACT-P total score:

Score range: 0-156

+ = = = FACT-P Total score
(PWB score) (SWB score) (EWB score) (FWB score) (PCS score)

# **Appendix 3: Scoring for PROMIS**

To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. In cases where individual items are skipped, the total raw scores can be prorated using the average of the raw scores of the complete items. This is acceptable as long as more than 50% of the items were answered at that specific visit. The prorated total raw scores with decimals should be rounded to the nearest whole number to translate to the corresponding T-score.

ARAMON V3.0 

The tables below are used to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.

| Fatigue 8a - Adult v1.0 | | |
|-----------------------------------|---------|-----|
| Short Form Conversion Table | | |
| Raw | Ticcoro | SE* |
| Score | T-score | 3E |
| 8 | 33.1 | 4.8 |
| 9 | 38.5 | 2.7 |
| 10 | 41.0 | 2.2 |
| 11 | 42.8 | 2.0 |
| 12 | 44.3 | 1.9 |
| 13 | 45.6 | 1.8 |
| 14 | 46.9 | 1.8 |
| 15 | 48.1 | 1.8 |
| 16 | 49.2 | 1.8 |
| 17 | 50.4 | 1.8 |
| 18 | 51.5 | 1.7 |
| 19 | 52.5 | 1.7 |
| 20 | 53.6 | 1.7 |
| 21 | 54.6 | 1.7 |
| 22 | 55.6 | 1.7 |
| 23 | 56.6 | 1.7 |
| 24 | 57.5 | 1.7 |
| 25 | 58.5 | 1.7 |
| 26 | 59.4 | 1.7 |
| 27 | 60.4 | 1.7 |
| 28 | 61.3 | 1.7 |
| 29 | 62.3 | 1.7 |
| 30 | 63.3 | 1.7 |
| 31 | 64.3 | 1.7 |
| 32 | 65.3 | 1.7 |
| 33 | 66.4 | 1.7 |
| 34 | 67.5 | 1.7 |
| 35 | 68.6 | 1.7 |
| 36 | 69.8 | 1.8 |
| 37 | 71.0 | 1.8 |
| 38 | 72.4 | 2.0 |
| 39 | 74.2 | 2.4 |
| 40 | 77.8 | 3.7 |
| *CE - Standard Error on T-score ! | | |

<sup>\*</sup>SE = Standard Error on T-score!

| A 1-16-0 | | 41 01 |
|---|---|---|
| Adult v2.0 – Physical Function 6b Short Form Conversion Table | | |
| Raw | Onn Conversion | Table |
| Summed<br>Score | T-score | SE* |
| 6 | 21.0 | 3.8 |
| 7 | 25.0 | 2.7 |
| 8 | 27.1 | 2.4 |
| 9 | 28.8 | 2.2 |
| 10 | 30.1 | 2.1 |
| 11 | 31.3 | 2.0 |
| 12 | 32.3 | 2.0 |
| 13 | 33.2 | 1.9 |
| 14 | 34.2 | 1.9 |
| 15 | 35.0 | 1.9 |
| 16 | 35.9 | 1.9 |
| 17 | 36.8 | 1.9 |
| 18 | 37.6 | 1.9 |
| 19 | 38.5 | 1.9 |
| 20 | 39.3 | 1.9 |
| 21 | 40.2 | 1.9 |
| 22 | 41.2 | 1.9 |
| 23 | 42.1 | 1.9 |
| 24 | 43.2 | 2.0 |
| 25 | 44.3 | 2.0 |
| 26 | 45.6 | 2.2 |
| 27 | 47.1 | 2.3 |
| 28 | 48.9 | 2.7 |
| 29 | 51.3 | 3.0 |
| 30 | 59.0 | 6.2 |
| *SE = Standar | d Error on T-sco | re metric |

PROMIS Physical Function 6b form

PROMIS Fatigue 8a form

ARAMON V3.0 

# Appendix 4: Randomized phase primary endpoint analysis for natural logarithm transformed Testosterone

Following data structure will be obtained for the Input dataset LN\_DATA. LN\_Change will be the difference between the LN(Testosterone) values at Visit 12 from the LN value at baseline.

```
Subjid trt LN_Change
Daro 0.5
Daro 0.9
ENZA 0.5
ENZA 0.8
```

The following SAS code will be used for the two-sample t-test.

```
PROC TTEST DATA=LN_DATA SIDES=2 ALPHA=0.05 H0=0;
CLASS TRT;
VAR LN_CHANGE;
RUN:
```

# Appendix 5: Lead-in phase analysis for natural logarithm transformed Testosterone and other endpoints using the log transformation

For the primary end point analysis, PROC TTEST procedure similar to Appendix 4: Randomized phase primary endpoint analysis for natural logarithm transformed Testosterone will be used without the CLASS statement.

For the lead-in phase, the following data structure will be obtained for the input dataset LN\_DATA to Proc Mixed. LN\_Change will be the difference between the LN(Testosterone) values at Visit from the LN value at baseline. During the lead-in phase there will be no enzalutamide data.

```
Subjid trt
           visit LN Change
          WK2 0.5
     Daro
     Daro WK4 0.9
     Daro
          WK8 1.3
     Daro
          WK16 1.6
          WK24 1.7
     Daro
     Daro WK36 1.7
     Daro
          Wk52 1.6
     Daro
          WK2 0.4
     Daro WK4 1.3
```

Following PROC Mixed code will be used.

```
PROC MIXED DATA = LN_DATA;
CLASS VISIT SUBJID;
```

ARAMON V3.0 

```
MODEL LN_CHANGE = VISIT /DDFM = KR;
RANDOM SUBJID;
REPEATED / TYPE = TOEP SUBJECT=SUBJID;
LSMEANS VISIT/ CL;
RUN;
```

Then the estimate for VISITS WK24 and WK52 will be retained. The dataset will have 2 lines. The fold change pair for each fold change (FC) can be computed as:

```
FC = EXP(Estimate);

LCL_FC = EXP(Estimate - StdErr*quantile('T', .975, DF));

UCL_FC = EXP(Estimate + StdErr*quantile('T', .975, DF));
```

These fold changes can be converted to Percent Change as:

```
PC = (FC-1)*100;

LCL_PC = (LCL_FC -1)*100;

UCL_PC = (UCL_FC -1)*100;
```

Similar code will be used for the other endpoints using the same transformation.

# Appendix 6: Randomized phase analysis for natural logarithm transformed Testosterone and other endpoints using the log transformation

The following data structure will be obtained for the input dataset LN\_DATA to Proc Mixed. LN\_Change will be the difference between the LN(Testosterone) values at Visit from the LN value at baseline.

```
Subjid trt
                LN Change
          visit
     Daro WK2 0.5
     Daro
          WK4 0.9
     Daro WK8 1.3
     Daro WK16 1.6
     Daro WK24 1.7
     Daro WK36 1.7
          Wk52 1.6
     Daro
     Daro WK2 0.4
     Daro WK4 1.3
     ENZA WK2 0.5
     ENZA WK4 2.2
     ENZA WK8 2.6
     ENZA WK16 2.8
```

The following PROC Mixed code will be used.

ARAMON V3.0 

```
PROC MIXED DATA = LN_DATA;
CLASS TRT VISIT SUBJID;
MODEL LN_CHANGE = TRT|VISIT /DDFM = KR;
RANDOM SUBJID(TRT);
REPEATED / TYPE = TOEP SUBJID(TRT);
LSMEANS TRT*VISIT/ DIFF SLICE = VISIT;
RUN;
```

Output the dataset created by LSMEANS. The data will be of the form:

| Obs | Effect | Trt | Visit | _Trt | _Visit | Estimate | StdErr | DF | t-value F | Probt |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | TRT*VISIT | Daro | WK2 | Daro | WK4 | 0.4 | 0.3 | XXX | XXX | 0.xx |
| 2 | TRT*VISIT | Daro | WK2 | Daro | WK8 | 0.8 | 0.32 | XXX | XXX | 0.xx |
| | TRT*VISIT | Daro | WK2 | ENZA | WK2 | -0.2 | 0.31 | XXX | xxx | 0.xx |
| | TRT*VISIT | Daro | WK52 | ENZA | WK52 | 0.4 | 0.3 | XXX | XXX | 0.xx |

From this dataset the records where 'Trt NE \_Trt', where Trt = 'Daro', where 'Visit = \_Visit' and Visit IN ('WK24','WK52") will be selected. This will select the two records where we are reporting results per the secondary objective. The fold change ratio (FCR) and the lower (LCL) and upper (UCL) confidence intervals for the fold change ratio will be obtained as:

```
FCR = EXP(Estimate);

LCL_FCR = EXP(Estimate - StdErr*quantile('T', .975, DF));

UCL_FCR = EXP(Estimate + StdErr*quantile('T', .975, DF))));
```

For fold change (FC) within treatment, the PROC MIXED will be repeated above with the following LSMEANS statement:

## LSMEANS TRT\*VISIT/CL;

Then the estimate for the Daro and ENZA for VISITS WK24 and WK52 will be retained. The dataset will have 6 lines. The fold change pair for each FCR can be computed as

```
FC = EXP(Estimate);

LCL_FC = EXP(Estimate - StdErr*quantile('T', .975, DF));

UCL_FC = EXP(Estimate + StdErr*quantile('T', .975, DF));
```

These fold changes can be converted to Percent Change as:

```
PC = (FC-1)*100;
LCL_PC = (LCL_FC -1)*100;
UCL_PC = (UCL_FC -1)*100;
```

Similar code can be used for the other endpoints using the same transformation.

ARAMON V3.0 

**Appendix 7: List of Abbreviations** 

| | ist of Addreviations |
|---|---|
| ADT | Androgen deprivation therapy |
| AE | Adverse event |
| AR | Androgen receptor |
| ARI | Androgen receptor inhibitor |
| BCR | Biochemical relapse |
| BMD | Bone mineral density |
| BSAP | Bone specific alkaline phosphatase |
| CI | Confidence interval |
| eCRF | Electronic case report form |
| CPET | Cardiopulmonary exercise test |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTX | C- Telopeptid |
| DEXA | Dual energy x-ray absorptiometry |
| DHT | Dihydrotestosterone |
| DHEA | Dehydroepiandrosterone |
| EC | Ethics committee |
| ECOG - PS | Eastern Cooperative Oncology Group Performance Status |
| eGFR | Estimated glomerular filtration rate |
| EOT | End of treatment |
| FACT-P | Functional Assessment of Cancer Therapy – Prostate Cancer |
| FAS | Full analysis set |
| FSH | Follicle-stimulating hormone |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation of Technical Requirements for |
| | Pharmaceuticals for Human Use |
| IRB | Institutional review board |
| ITT | Intent-to-treat |
| IWRS | Interactive web randomization system |
| LH | luteinizing hormone |
| LPLT | Last participant last treatment |
| LPLV | Last participant last visit |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| NCI - CTCAE | National Cancer Institute-Common Terminology Criteria for Adverse Events |
| PROMIS | Participant reported outcome measurement information system |
| PSA | Prostate-specific antigen |
| PSADT | PSA doubling time |
| PT | Preferred term |
| QOL | Quality of life |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| TSH | Thyroid stimulating hormone |
| SHBG | Sex hormone binding globulin |

| CONFIDENTIAL | Statistical Analysis Plan |
|--------------|---------------------------|
| | 1841788 / 21953 |

ARAMON V3.0 

| TEAE | Treatment emergent adverse events |
|-------|-------------------------------------------|
| TESAE | Treatment emergent serious adverse events |